CLINICAL TRIAL: NCT02205359
Title: AdaptResponse Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AdaptResponse
Record Dates: First submitted 2014-07-18; First posted 2014-07-31 (Estimated); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure With Left Bundle Branch Block
Keywords: AdaptivCRT; aCRT

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aCRT ON (Experimental): The aCRT algorithm has been developed to provide RV-synchronized LV pacing when intrinsic AV conduction is normal or BiV pacing otherwise
  Interventions: Device: aCRT ON
- aCRT OFF (Active Comparator): Standard CRT
  Interventions: Device: aCRT OFF

INTERVENTIONS:
Device: aCRT ON — CRT device with AdaptivCRT enabled (AdaptivBiV and LV)
  Arms: aCRT ON
Device: aCRT OFF — CRT device with AdaptivCRT disabled
  Arms: aCRT OFF

SUMMARY:
The purpose of this clinical study is to test the hypothesis that market released Cardiac Resynchronization Therapy (CRT) devices which contain the AdaptivCRT® (aCRT) algorithm have a superior outcome compared to standard CRT devices in CRT indicated patients with normal atrio-ventricular (AV) conduction and left bundle branch block (LBBB).

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to sign and date the study Patient Informed Consent Form.
* Subject is indicated for a CRT device according to local guidelines.
* Sinus Rhythm at time of enrollment
* Complete Left Bundle Branch Block (LBBB) as documented on an ECG (within 30 days prior to enrollment). Strauss Criteria used for LBBB.
* Intrinsic, normal AV conduction as documented on an ECG by a PR interval less than or equal to 200ms (within 30 days prior to enrollment).
* Left ventricular ejection fraction less than or equal to 35% (documented within 180 days prior to enrollment).
* NYHA class II, III or IV (documented within 30 days prior to enrollment) despite optimal medical therapy. Optimal medical therapy is defined as maximal tolerated dose of Beta-blockers and a therapeutic dose of ACE-I, ARB or Aldosterone Antagonist.

Exclusion Criteria:

* Subject is less than 18 years of age (or has not reached minimum age per local law).
* Subject is not expected to remain available for at least 2 years of follow-up visits.
* Subject has permanent atrial arrhythmias for which pharmacological therapy and/or cardioversion have been unsuccessful or have not been attempted
* Subject is, or previously has been, receiving cardiac resynchronization therapy.
* Subject is currently enrolled or planning to participate in a potentially confounding drug or device trial during the course of this study. Co-enrollment in concurrent trials is only allowed when documented pre-approval is obtained from the Medtronic study manager.
* Subject has unstable angina, or experienced an acute myocardial infarction (MI) or received coronary artery revascularization (CABG) or coronary angioplasty (PTCA) within 30 days prior to enrollment.
* Subject has a mechanical tricuspid heart valve or is scheduled to undergo valve repair or valve replacement during the course of the study.
* Subject is post heart transplant (subjects on the heart transplant list for the first time are not excluded).
* Subject has a limited life expectancy due to non-cardiac causes that would not allow completion of the study.
* Subject is pregnant (if required by local law, women of child-bearing potential must undergo a pregnancy test within seven days prior to device implant).
* Subject meets any exclusion criteria required by local law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3797 (Actual)
Dates: Start 2014-08; Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Wilkoff, MD, Study Chair — The Cleveland Clinic
Locations (220):
- United States (90):
  - CardioVascular Associates of Mesa, Mesa, Arizona
  - Phoenix Cardiovascular Research Group, LLC, Phoenix, Arizona
  - Saint Vincent Heart Clinic Arkansas, Little Rock, Arkansas
  - Scripps Green Hospital Scripps Clinic Torrey Pines, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Coggins & Levy Medical Associates, San Jose, California
  - Stanford Hospital & Clinics, Stanford, California
  - Saint Joseph's Medical Center, Stockton, California
  - Penrose Hospital, Colorado Springs, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Heart & Vascular Institute of Florida, Clearwater, Florida
  - Florida Heart Rhythm Specialists PLLC, Fort Lauderdale, Florida
  - The Cardiac & Vascular Institute, Gainesville, Florida
  - First Coast Cardiovascular Institute PA, Jacksonville, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - AdventHealth Cardiovascular Research Institute, Orlando, Florida
  - Cardiology Institute of Northwest Florida, Panama City, Florida
  - University of South Florida Health (USF), Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northwerstern University, Chicago, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Saint Francis Medical Group Indiana Heart Physician, Indianapolis, Indiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - MedStar Health Research Institute, Baltimore, Maryland
  - Massachusetts General Hospital (Boston MA), Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - North Memorial Heart and Vascular Institute, Robbinsdale, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Mid America Heart Institute (MAHI), Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Glacier View Research Institute Cardiology, Kalispell, Montana
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - New York Methodist Hospital, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Central New York Cardiology, Utica, New York
  - Asheville Cardiology Associate PA, Asheville, North Carolina
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - Wake Forest Baptist Health High Point Medical Center, High Point, North Carolina
  - Raleigh Cardiology Associates, Raleigh, North Carolina
  - Bethesda North Hospital, Cincinnati, Ohio
  - The Lindner Research Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Mount Carmel East, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - North Ohio Heart-Elyria, Elyria, Ohio
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - Sacred Heart Medical Center, Eugene, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Capital Area Research, Camp Hill, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Mercer Bucks Cardiology, Newtown, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Great Valley Cardiology, Scranton, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Sutherland Cardiology Clinic, Memphis, Tennessee
  - Centennial Heart Cardiovascular Consultants LLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - The University of Texas (UT) Southwestern Medical Center, Dallas, Texas
  - CHI St. Luke's Heath Baylor College of Medicine Medical Center, Houston, Texas
  - Baylor Research Institute, Plano, Texas
  - EP Heart LLC, The Woodlands, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - The University of Vermont Medical Center Inc, Burlington, Vermont
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Cardiovascular Specialists PC, Richmond, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Swedish Medical Center Cherry Hill, Seattle, Washington
  - Providence Spokane Cardiology, Spokane, Washington
  - CAMC Health Education & Research Institute Inc, Charleston, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- Australia (4):
  - John Hunter Hospital, New Lambton, New South Wales
  - Austin Hospital, Heidelberg, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Saint Vincent's Hospital (Sydney), Sydney
- Austria (2):
  - Landeskrankenhaus Innsbruck - Universitätskliniken, Innsbruck
  - Allgemeines Krankenhaus der Stadt Linz, Linz
- Belgium (2):
  - AZ Sint-Jan Brugge-Oostende av, Bruges
  - Ziekenhuis Oost Limburg - Campus St.-Jan, Genk
- Canada (7):
  - London Health Sciences Centre - University Campus, London
  - McGill Universtiy Health Centre (MUHC), Montreal
  - Southlake Regional Health Centre, Newmarket
  - University of Ottawa Heart Institute, Ottawa
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec
  - Royal Columbian Hospital, Vancouver
  - Vancouver General Hospital, Vancouver
- Odense Universitetshospital, Odense C, Denmark
- Finland (2):
  - Keski-Suomen Keskussairaala, Jyväskylä
  - Satakunnan keskussairaala, Pori
- France (17):
  - Centre Hospitalier Universitaire de Amiens - Hôpital SU, Amiens
  - CHRU Tours - Hôpital Trousseau, Chambray-lès-Tours
  - Centre Hospitalier Universitaire de Clermont-Ferrand - Gabriel-Montpied, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHRU La Rochelle, La Rochelle
  - Centre Hospitalier Universitaire de Grenoble-Hopital Albert Michallon, La Tronche
  - CHRU de Lille, Lille
  - groupe Hospitalier de L'Institut Catholique de Lille - Hôpital Saint-Philibert, Lomme
  - Hopital prive Clairval - Ramsay Sante, Marseille
  - Hôpital de la Timone - Centre Hospitalier Universitaire de Marseille, Marseille
  - Institut Hospitalier Jacques Cartier, Massy
  - CHR Metz-Thionville Hôpital de Mercy, Metz
  - CHRU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - Nouvelles Cliniques Nantaises, Nantes
  - CMC-Clinique Ambroise Pare, Neuilly-sur-Seine
  - Hôpital Pontchaillou - CHU de Rennes, Rennes
  - CHU Toulouse - Hôpital Rangueil, Toulouse
- Germany (17):
  - Immanuel Diakonie Group - Evangelisch-Freikirchlichen Krankenhaus und Herzzentrum Brandenburg, Bernau bei Berlin
  - Herz- und Diabeteszentrum NRW - Ruhr-Universität Bochum, Bochum
  - MVZ am Küchwald GmbH ambulantes Herz Zentrum Chemnitz, Chemnitz
  - Klinikum Coburg GmbH, Coburg
  - Praxisklinik Herz und Gefässe - Akademische Lehrpraxisklinik der TU Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätskliniken des Saarlandes, Homburg/Saar
  - Universitätsklinikum Jena - Friedrich Schiller Universität, Jena
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - Märkische Gesundheitsholding GmbH & Co. KG - Klinikum Lüdenscheid, Lüdenscheid
  - Berufsgenossenschaftliche Universitätsklinik Bergmannsheil GmbH, Lüdenscheid
  - Otto von Guericke Universität - Universitätsklinikum Magdeburg A.ö.R., Magdeburg
  - Kliniken Maria Hilf GmbH Mönchengladbach - Krankenhaus St. Franziskus, Mönchengladbach
  - Klinikum der Universität München - Campus Großhadern, München
  - Herz Riesa, Gemeinschaftspraxis, Riesa
  - Universitätsklinikum Ulm, Ulm
- Hungary (2):
  - Magyar Honvédség Honvédkorház, Budapest
  - Semmelweis Egyetem AOK, Budapest
- India (2):
  - Medanta - The Medicity, Gūrgaon
  - Fortis Escorts Heart Institute, New Delhi
- Italy (6):
  - Policlinico Sant' Orsola - Malpighi, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Ospedale Civile Madonna Della Navicella, Chioggia
  - Azienda Ospedaliera Carlo Poma, Mantova
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (10):
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Chiba University Hospital, Chiba
  - Kokura Memorial Hospital, Kitakyushu
  - Kyorin University Hospital, Mitaka-Shi
  - Nagoya University Hospital, Nagoya
  - Sakakibara Heart Institute of Okayama, Okayama
  - Saitama Medical Center Jichi Medical University, Shimonoseki-Shi
  - National Cerebral and Cardiovascular Center, Suita-Shi
  - Fujita Health University Hospital, Toyoake
  - University of Fukui Hospital, Tsukuba
- Hospital Angeles Leon, León, Guanajuato, Mexico
- Netherlands (8):
  - Academisch Medisch Centrum, Amsterdam
  - Amphia Ziekenhuis - Locatie Molengracht Breda, Breda
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Canisius-Wilhelmina ziekenhuis, Nijmegen
  - Maasstad Ziekenhuis, Rotterdam
  - Erasmus Medisch Centrum, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Isala Klinieken - Locatie Weezenlanden, Zwolle
- Helse Bergen HF - Haukeland Universitetssjukehus, Bergen, Norway
- Poland (6):
  - Wojewódzki Szpital Zespolony im. Ludwika Perzyny w Kaliszu, Kalisz
  - Górnośląskie Centrum Medyczne im prof Leszka Gieca Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Regional Hospital Szpital Wojewodski, Kielce
  - Wojewódzki Szpital Specjalistyczny im. Stefana Kardynała Wyszyńskiego, Lublin
  - Spital Wojewodzki nr 2, Rzeszów
  - Slaskie Centrum Chorob Serca, Zabrze
- Portugal (3):
  - Unidade Local de Saude do Baixo Alentejo, EPE - Hospital José Joaquim Fernandes, Beja
  - Centro Hospitalar de Coimbra, Coimbra
  - Hospital de Espírito Santo E.P.E., Evora
- Puerto Rico (2):
  - The Arrhythmia Group, Coto Laurel
  - Cardiovascular Center, San Juan
- Russia (3):
  - AV Vishnevsky Institute of Surgery of the Ministry of Health of the Russian Federation, Moscow
  - EN Meshalkin National medical research center of the Ministry of Health of the Russian Federation, Novosibirsk
  - Almazov National Medical Research Centre, Saint Petersburg
- Saudi Arabia (4):
  - King Abdul Aziz University Hospital, Jeddah
  - King Fahad Armed Forces Hospital, Jeddah
  - King Faisal Specialist Hospital & Research Center, Riyadh
  - The College of Medicine & King Khalid University Hospital, King Saud University, Riyadh
- Slovakia (2):
  - Stredoslovensky ustav srdcovych a cievnych chorob a.s, Banská Bystrica
  - NUSCH, a.s., Bratislava
- South Korea (6):
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (10):
  - Hospital Universitario Infanta Cristina, Badajoz
  - Nuevo Hospital de Burgos, Burgos
  - Hospital Virgen de la Arrixaca, El Palmar
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Clínico Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocío, Seville
  - Complexo Hospitalario Universitario de Vigo - Hospital Xeral Cíes, Vigo
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (2):
  - Karolinska Universitetssjukhuset, Solna
  - Akademiska Sjukhuset, Uppsala
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - HFR Fribourg - Hôpital cantonal, Fribourg
  - Kantonsspital St.Gallen, Sankt Gallen
- Taiwan (2):
  - National Taiwan University Hospital Hsin Chu Branch, Hsinchu
  - National Taiwan University Hospital, Taipei
- United Kingdom (5):
  - Golden Jubilee National Hospital - NHS Trust, Glasgow
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - University Hospitals of North Midlands NHS Trust - Royal Stoke University Hospital, Liverpool
  - Royal Brompton & Harefield NHS Foundation Trust - Royal Brompton Hospital, London
  - Manchester University NHS Foundation Trust - Wythenshawe Hospital, Manchester

REFERENCES:
- [Derived] Wilkoff BL, Filippatos G, Leclercq C, Gold MR, Hersi AS, Kusano K, Mullens W, Felker GM, Kantipudi C, El-Chami MF, Essebag V, Pierre B, Philippon F, Perez-Gil F, Chung ES, Sotomonte J, Tung S, Singh B, Bozorgnia B, Goel S, Ebert HH, Varma N, Quan KJ, Salerno F, Gerritse B, van Wel J, Schaber DE, Fagan DH, Birnie D; AdaptResponse investigators. Adaptive versus conventional cardiac resynchronisation therapy in patients with heart failure (AdaptResponse): a global, prospective, randomised controlled trial. Lancet. 2023 Sep 30;402(10408):1147-1157. doi: 10.1016/S0140-6736(23)00912-1. Epub 2023 Aug 24. PMID 37634520
- [Derived] Wilkoff BL, Birnie D, Gold MR, Hersi AS, Jacobs S, Gerritse B, Kusano K, Leclercq C, Mullens W, Filippatos G. Differences in clinical characteristics and reported quality of life of men and women undergoing cardiac resynchronization therapy. ESC Heart Fail. 2020 Oct;7(5):2972-2982. doi: 10.1002/ehf2.12914. Epub 2020 Aug 13. PMID 32790108
- [Derived] Filippatos G, Birnie D, Gold MR, Gerritse B, Hersi A, Jacobs S, Kusano K, Leclercq C, Mullens W, Wilkoff BL; AdaptResponse Investigators. Rationale and design of the AdaptResponse trial: a prospective randomized study of cardiac resynchronization therapy with preferential adaptive left ventricular-only pacing. Eur J Heart Fail. 2017 Jul;19(7):950-957. doi: 10.1002/ejhf.895. PMID 28708290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between August 2014 and January 2019
Pre-assignment Details: After subject enrollment, subjects were first implanted with a Medtronic device compatible with the AdaptivCRT algorithm. After successful implant subjects were randomized.
Groups:
- aCRT ON: The AdaptivCRT (aCRT) algorithm has been developed to provide RV-synchronized LV pacing when intrinsic AV conduction is normal or BiV pacing otherwise
  aCRT ON: CRT device with AdaptivCRT enabled (AdaptivBiV and LV)
- aCRT OFF: Standard CRT
  aCRT OFF: CRT device programmed to Nonadaptive CRT
Period: Overall Study
Arm/Group | aCRT ON | aCRT OFF
Started (Number of subjects following successful implant and randomization) | 1810 | 1807
Completed | 1117 | 1096
Not Completed | 693 | 711
Not completed — Death | 293 | 327
Not completed — Lost to Follow-up | 182 | 162
Not completed — Physician Decision | 51 | 53
Not completed — Withdrawal by Subject | 167 | 169

BASELINE CHARACTERISTICS:
Population: Number of subjects randomized following successful implant
Groups:
- Total: Total of all reporting groups
Arm/Group | aCRT ON | aCRT OFF | Total
Number analyzed (Participants) | 1810 | 1807 | 3617
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (11.1) | 65.2 (11.0) | 64.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 782 | 786 | 1568
  Male | 1028 | 1021 | 2049
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
NYHA class [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification, places patients in one of four categories based on limitations of physical activity.
  The categories are as follows:
  I: No limitation of physical activity. II: Slight limitation of physical activity. Comfortable at rest. III: Marked limitation of physical activity. Comfortable at rest. IV: Symptoms of heart failure at rest. Any physical activity causes further discomfort.
  Participants
    NYHA class II | 881 | 867 | 1748
    NYHA class III | 908 | 912 | 1820
    NYHA class IV | 21 | 28 | 49

OUTCOME MEASURES:

1. Primary Outcome: Combined Endpoint of All-cause Mortality and Intervention for Heart Failure Decompensation
Description: The first occurrence of death or intervention for heart failure decompensation (defined as an event requiring invasive intervention or inpatient hospitalization).
Time Frame: from subject randomization until the first occurrence of death or intervention for heart failure decompensation, median follow-up 4.9 years (max. follow-up 8.1 years)
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Groups:
- aCRT ON: The aCRT algorithm has been developed to provide RV-synchronized LV pacing when intrinsic AV conduction is normal or BiV pacing otherwise
  aCRT ON: CRT device with AdaptivCRT enabled
Arm/Group | aCRT ON | aCRT OFF
Number analyzed (Participants) | 1810 | 1807
Participants | 430 | 470
Statistical Analysis 1: Comparison: aCRT ON vs aCRT OFF; Test type: Superiority; p = 0.077, Regression, Cox; Stratified by NYHA class and with investigational site as a random effect; Hazard Ratio (HR) = 0.888, 95% CI 2-sided [0.779 to 1.013], Standard Error of Mean 0.067 — Stratified by NYHA class and with investigational site as a random effect, Standard Error reported on log hazard scale

2. Secondary Outcome: All-cause Mortality
Description: All-cause mortality in the aCRT ON group vs the aCRT OFF group
Time Frame: from subject randomization until the occurrence of death, median follow-up 4.9 years (max. follow-up 8.1 years)
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | aCRT ON | aCRT OFF
Number analyzed (Participants) | 1810 | 1807
Participants | 293 | 327
Statistical Analysis 1: Comparison: aCRT ON vs aCRT OFF; Test type: Superiority; p = 0.12, Regression, Cox; Stratified by NYHA class and with investigational site as a random effect; Hazard Ratio (HR) = 0.881, 95% CI 2-sided [0.752 to 1.032], Standard Error of Mean 0.081 — Stratified by NYHA class and with investigational site as a random effect, Standard Error reported on log hazard scale

3. Secondary Outcome: Percent of Patients With Interventions for Heart Failure Decompensation
Description: First occurence of intervention for heart failure decompensation is defined as an event requiring invasive intervention or inpatient hospitalization.
Time Frame: from subject randomization until the first occurrence of intervention for heart failure decompensation, median follow-up 4.9 years (max. follow-up 8.1 years)
Population: all randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | aCRT ON | aCRT OFF
Number analyzed (Participants) | 1810 | 1807
Participants | 238 | 255
Statistical Analysis 1: Comparison: aCRT ON vs aCRT OFF; Test type: Superiority; p = 0.28, Regression, Cox; Stratified by NYHA class and with investigational site as a random effect; Hazard Ratio (HR) = 0.906, 95% CI 2-sided [0.759 to 1.082], Standard Error of Mean 0.090 — Stratified by NYHA class and with investigational site as a random effect, Standard Error reported on log hazard scale

4. Secondary Outcome: Clinical Composite Score
Description: The Clinical Composite Score (CCS) classifies patients according their clinical status at 6 months post randomization into categories Improved, Unchanged, and Worsened. A patient is classified Worsened in case of death, hospitalization for worsening heart failure, worsened NYHA class (using last observation carried forward), or worsened status on the Global Assessment Score. Also patients that exit the study or cross over because of worsening heart failure are classified Worsened. A patient is classified Improved when not Worsened and there is an improvement in NYHA class or Global Assessment Score. Patients that are not Worsened or Improved are Unchanged.
Time Frame: CCS at 6 month post randomization
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | aCRT ON | aCRT OFF
Number analyzed (Participants) | 1810 | 1807
Participants
  Improved | 1250 | 1291
  Unchanged | 422 | 387
  Worsened | 138 | 129
Statistical Analysis 1: Comparison: aCRT ON vs aCRT OFF; Test type: Superiority — Endpoint for statistical analysis is the proportion Improved; p = 0.11, Regression, Logistic; Stratified by NYHA class and with investigational site as a random effect; Odds Ratio (OR) = 0.888, 95% CI 2-sided [0.768 to 1.026], Standard Error of Mean 0.074 — Standard Error is on log-odds ratio scale

5. Secondary Outcome: Atrial Fibrillation
Description: Occurrence of atrial fibrillation lasting >6 hours in one day
Time Frame: from subject randomization until the first occurrence of atrial fibrillation lasting >6 hours in one day, median follow-up 4.9 years (max. follow-up 8.1 years)
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | aCRT ON | aCRT OFF
Number analyzed (Participants) | 1810 | 1807
Participants | 317 | 316
Statistical Analysis 1: Comparison: aCRT ON vs aCRT OFF; Test type: Superiority; p = 0.89, Regression, Cox; Stratified by NYHA class and with investigational site as a random effect; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.85 to 1.16]

6. Secondary Outcome: Change in Quality of Life Measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The overall summary score of the Kansas City Cardiomyopathy Questionnaire will be analyzed. The KCCQ measures Quality of Life on a 0-100 scale with higher scores indicating better QoL
Time Frame: from baseline to 24M follow up
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | aCRT ON | aCRT OFF
Number analyzed (Participants) | 1810 | 1807
score on a scale
  Overall summary score mean at 24M | 80.3 (19.7) | 81.8 (19.0)
  Overall summary score change from baseline to 24M | 16.8 (21.2) | 16.5 (20.4)
Statistical Analysis 1: Comparison: aCRT ON vs aCRT OFF; Test type: Superiority; p = 0.88, ANCOVA; Stratified by NYHA class and with investigational site as a random effect; Difference in mean change from baseline = -0.07, 95% CI 2-sided [-1.03 to 0.89]

7. Secondary Outcome: Change in Quality of Life Measured by the EQ-5D
Description: The EQ-5D descriptive system comprises the following five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN /DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has three levels: no problems, some problems, extreme problems (labelled 1-3). We calculated the EQ-5D summary index by applying a specific formula providing a valuation to the health states (Shaw et al. Medical Care 2005). For the summary index, value 0 represents health that is valued as equal to death and value 1 represents best possible health.
Time Frame: from baseline to 24M follow up
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | aCRT ON | aCRT OFF
Number analyzed (Participants) | 1810 | 1807
score on a scale
  Mean index score at 24M | 0.848 (0.173) | 0.862 (0.173)
  Mean index score change from baseline to 24M | 0.054 (0.190) | 0.048 (0.180)
Statistical Analysis 1: Comparison: aCRT ON vs aCRT OFF; Test type: Superiority; p = 0.75, ANCOVA; Stratified by NYHA class and with investigational site as a random effect; Difference in mean change from baseline = 0.0013, 95% CI 2-sided [-0.0068 to 0.0094]

8. Secondary Outcome: All-cause Re-admissions Within 30 Days After a Heart Failure Admission Per 100 Patient Years
Description: All-cause hospital re-admissions within 30 days after discharge from a heart failure admission are reported as number of cases per 100 patient years
Time Frame: from subject randomization until study exit, median follow-up 4.9 years (max. follow-up 8.1 years)
Population: All randomized subjects
Measure: Number; unit: readmissions per 100 patient years
Arm/Group | aCRT ON | aCRT OFF
Number analyzed (Participants) | 1810 | 1807
readmissions per 100 patient years | 1.07 | 0.93
Statistical Analysis 1: Comparison: aCRT ON vs aCRT OFF; Test type: Superiority; p = 0.52, negative binomial regression; Stratified by NYHA class; rate ratio = 1.15, 95% CI 2-sided [0.75 to 1.75]

ADVERSE EVENTS:
Time Frame: the data were collected from subject randomization until death or study completion, median follow-up 4.9 years (maximum follow-up 8.1 years)
Description: The clinical study collected all serious and all system, procedure, and/or cardiovascular related adverse events. Healthcare Utilizations where these AEs occurred were also collected. The Endpoint Adjudication Committee reviewed all applicable Healthcare Utilizations and all study reportable events during the study, assessing outpatient treatment and hospitalizations, to determine HF relatedness and AF relatedness for the study objectives.
Arm/Group | aCRT ON | aCRT OFF
All-Cause Mortality (participants affected / at risk) | 293/1810 | 327/1807
Serious Adverse Events (participants affected / at risk) | 1072/1810 | 1073/1807
Other Adverse Events (participants affected / at risk) | 773/1810 | 785/1807
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | aCRT ON (N=1810) | aCRT OFF (N=1807)
Anaemia (Blood and lymphatic system disorders) | 41 (50) | 47 (50)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 3 (3) | 7 (7)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Idiopathic CD4 lymphocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 (5) | 13 (14)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Accelerated idioventricular rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 9 (10) | 5 (5)
Acute left ventricular failure (Cardiac disorders) | 41 (55) | 42 (50)
Acute myocardial infarction (Cardiac disorders) | 31 (39) | 42 (42)
Angina pectoris (Cardiac disorders) | 28 (29) | 23 (24)
Angina unstable (Cardiac disorders) | 9 (12) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 3 (3) | 5 (5)
Arrhythmia (Cardiac disorders) | 1 (1) | 6 (6)
Arrhythmia supraventricular (Cardiac disorders) | 3 (3) | 2 (2)
Arrhythmic storm (Cardiac disorders) | 6 (7) | 5 (6)
Arteriosclerosis coronary artery (Cardiac disorders) | 3 (3) | 3 (3)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 136 (183) | 154 (202)
Atrial flutter (Cardiac disorders) | 20 (26) | 24 (29)
Atrial tachycardia (Cardiac disorders) | 4 (4) | 7 (7)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 4 (4)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 30 (31) | 19 (20)
Cardiac asthma (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 206 (305) | 242 (396)
Cardiac failure acute (Cardiac disorders) | 41 (55) | 55 (67)
Cardiac failure chronic (Cardiac disorders) | 26 (34) | 26 (26)
Cardiac failure congestive (Cardiac disorders) | 86 (144) | 76 (112)
Cardiac flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac perforation (Cardiac disorders) | 3 (3) | 6 (6)
Cardiac sarcoidosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 2 (2) | 5 (5)
Cardio-respiratory arrest (Cardiac disorders) | 4 (4) | 4 (4)
Cardiogenic shock (Cardiac disorders) | 21 (22) | 22 (25)
Cardiomegaly (Cardiac disorders) | 3 (3) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 6 (6) | 4 (4)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 4 (5) | 9 (9)
Chronic left ventricular failure (Cardiac disorders) | 7 (8) | 4 (5)
Congestive cardiomyopathy (Cardiac disorders) | 4 (7) | 3 (4)
Coronary artery disease (Cardiac disorders) | 22 (23) | 24 (29)
Coronary artery occlusion (Cardiac disorders) | 3 (3) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 4 (4) | 7 (7)
Coronary ostial stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary vein stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Heart valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac mass (Cardiac disorders) | 2 (2) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 5 (8) | 3 (3)
Left ventricular dilatation (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 8 (8) | 6 (6)
Mitral valve incompetence (Cardiac disorders) | 13 (16) | 21 (22)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 6 (6) | 4 (4)
Myocardial injury (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 7 (7) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 19 (19) | 20 (21)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 7 (8) | 5 (6)
Pericarditis constrictive (Cardiac disorders) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 2 (2)
Right ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 3 (3)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 12 (13) | 13 (14)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 3 (3)
Tachycardia (Cardiac disorders) | 10 (11) | 11 (11)
Torsade de pointes (Cardiac disorders) | 2 (2) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 2 (2) | 4 (4)
Tricuspid valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 4 (4)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular dyssynchrony (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 13 (14) | 17 (19)
Ventricular fibrillation (Cardiac disorders) | 24 (27) | 25 (29)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 87 (127) | 92 (137)
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Congenital cardiovascular anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Myocardial bridging (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear canal stenosis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 3 (3)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 2 (2)
Cushing's syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Parathyroid disorder (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 4 (4) | 0 (0)
Thyrotoxic crisis (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 8 (10) | 5 (6)
Choroidal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Entropion (Eye disorders) | 1 (1) | 0 (0)
Epiretinal membrane (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 2 (2)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 10 (12)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 4 (4)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 4 (4)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 5 (5) | 5 (5)
Colitis ischaemic (Gastrointestinal disorders) | 3 (3) | 3 (3)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 8 (9)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 (1) | 1 (2)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 3 (3) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal varices (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (2)
Enteritis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 22 (25) | 24 (25)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 3 (3) | 4 (4)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 8 (8) | 6 (6)
Intestinal angina (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 4 (4) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 3 (4)
Oesophageal achalasia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 1 (2) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 4 (5) | 5 (5)
Pancreatitis acute (Gastrointestinal disorders) | 6 (8) | 3 (3)
Pancreatitis chronic (Gastrointestinal disorders) | 2 (2) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Proctitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 6 (6) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 6 (6) | 6 (7)
Small intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 5 (5) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4) | 3 (3)
Volvulus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Volvulus of small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Adverse drug reaction (General disorders) | 3 (3) | 1 (1)
Asthenia (General disorders) | 6 (6) | 5 (5)
Chest discomfort (General disorders) | 3 (3) | 1 (1)
Chest pain (General disorders) | 28 (33) | 20 (30)
Complication associated with device (General disorders) | 0 (0) | 1 (2)
Cyst (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 47 (47) | 45 (45)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 3 (3) | 1 (1)
General physical health deterioration (General disorders) | 2 (3) | 1 (1)
Generalised oedema (General disorders) | 2 (2) | 0 (0)
Hernia (General disorders) | 1 (1) | 2 (2)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 1 (1)
Implant site dehiscence (General disorders) | 1 (1) | 1 (1)
Implant site extravasation (General disorders) | 1 (1) | 0 (0)
Implant site haematoma (General disorders) | 8 (8) | 5 (5)
Implant site haemorrhage (General disorders) | 3 (3) | 0 (0)
Implant site pain (General disorders) | 9 (9) | 2 (2)
Implant site swelling (General disorders) | 0 (0) | 1 (1)
Implant site ulcer (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 2 (2) | 0 (0)
Medical device site calcification (General disorders) | 0 (0) | 1 (1)
Medical device site discharge (General disorders) | 1 (1) | 0 (0)
Medical device site extravasation (General disorders) | 1 (1) | 0 (0)
Medical device site haemorrhage (General disorders) | 0 (0) | 1 (1)
Medical device site irritation (General disorders) | 1 (1) | 0 (0)
Medical device site mass (General disorders) | 1 (1) | 0 (0)
Medical device site pain (General disorders) | 1 (1) | 1 (1)
Multimorbidity (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 6 (6) | 5 (5)
Necrosis (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 22 (32) | 20 (22)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 5 (6) | 3 (3)
Organ failure (General disorders) | 1 (1) | 0 (0)
Pacemaker generated arrhythmia (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (2)
Pelvic mass (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 1 (1)
Phantom shocks (General disorders) | 1 (1) | 1 (1)
Physical deconditioning (General disorders) | 1 (1) | 0 (0)
Prosthetic cardiac valve stenosis (General disorders) | 0 (0) | 1 (1)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 1 (1)
Stent-graft endoleak (General disorders) | 2 (2) | 0 (0)
Sudden cardiac death (General disorders) | 5 (5) | 5 (5)
Sudden death (General disorders) | 1 (1) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 4 (4)
Unevaluable event (General disorders) | 2 (2) | 1 (1)
Vascular stent stenosis (General disorders) | 2 (2) | 0 (0)
Vascular stent thrombosis (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 2 (3)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary-bronchial fistula (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 5 (5) | 5 (5)
Cholecystitis acute (Hepatobiliary disorders) | 8 (8) | 10 (10)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 9 (9) | 8 (9)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Congestive hepatopathy (Hepatobiliary disorders) | 1 (1) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (2) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 2 (3)
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 1 (1) | 1 (1)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Heart transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1)
Solid organ transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 4 (4)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 4 (4) | 3 (3)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 5 (5)
Arteriovenous fistula site infection (Infections and infestations) | 1 (1) | 0 (0)
Arteriovenous graft site infection (Infections and infestations) | 1 (2) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 7 (8) | 5 (5)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 11 (13) | 12 (13)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 18 (18) | 22 (22)
COVID-19 pneumonia (Infections and infestations) | 23 (23) | 17 (17)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 2 (4) | 0 (0)
Cellulitis (Infections and infestations) | 18 (19) | 14 (14)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Chest wall abscess (Infections and infestations) | 0 (0) | 2 (2)
Chronic sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Citrobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 5 (7) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 5 (6) | 6 (6)
Coccidioidomycosis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 6 (6) | 4 (5)
Dermo-hypodermitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 4 (5) | 9 (10)
Device related sepsis (Infections and infestations) | 2 (2) | 1 (1)
Diabetic foot infection (Infections and infestations) | 3 (3) | 1 (1)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Disseminated coccidioidomycosis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 5 (5) | 9 (10)
Diverticulitis intestinal perforated (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 6 (6) | 12 (12)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 3 (3) | 3 (3)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1)
Fournier's gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 2 (2) | 3 (4)
Gas gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (7) | 6 (6)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 1 (1) | 0 (0)
Implant site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 14 (14) | 5 (6)
Infection (Infections and infestations) | 3 (3) | 3 (3)
Infection susceptibility increased (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 10 (10) | 8 (8)
Infusion site infection (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 2 (2)
Intestinal sepsis (Infections and infestations) | 0 (0) | 2 (2)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 3 (3)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Norovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 8 (10) | 6 (7)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 4 (5) | 2 (2)
Pneumonia (Infections and infestations) | 84 (105) | 80 (93)
Pneumonia aspiration (Infections and infestations) | 7 (8) | 5 (5)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 5 (5) | 3 (3)
Pyelonephritis (Infections and infestations) | 5 (5) | 8 (8)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 5 (5)
Rhinovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Salmonella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 30 (31) | 39 (50)
Septic shock (Infections and infestations) | 26 (27) | 17 (17)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 10 (10)
Staphylococcal infection (Infections and infestations) | 4 (5) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 1 (1)
Urinary tract infection (Infections and infestations) | 35 (51) | 50 (57)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 7 (7) | 16 (16)
Vascular device infection (Infections and infestations) | 2 (2) | 3 (3)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulval cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 2 (2)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Anastomotic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Aortic pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula maturation failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac vein dissection (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cardiac vein perforation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary bypass stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Device use issue (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 7 (8) | 4 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Femur fracture (Injury, poisoning and procedural complications) | 7 (7) | 6 (6)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 7 (8) | 9 (10)
Humerus fracture (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 2 (4) | 1 (1)
Pocket erosion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Post procedural hypotension (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Shunt stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spleen contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Twiddler's syndrome (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access steal syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Anticoagulation drug level above therapeutic (Investigations) | 2 (2) | 1 (2)
Anticoagulation drug level below therapeutic (Investigations) | 1 (1) | 0 (0)
Arthroscopy (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Blood pressure orthostatic abnormal (Investigations) | 1 (1) | 0 (0)
Catheterisation cardiac (Investigations) | 2 (2) | 0 (0)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (1)
Escherichia test positive (Investigations) | 1 (1) | 0 (0)
Gram stain positive (Investigations) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1)
Heart rate decreased (Investigations) | 1 (1) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Influenza B virus test positive (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1)
Myocardial necrosis marker increased (Investigations) | 1 (1) | 0 (0)
Streptococcus test positive (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 3 (3) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 13 (15) | 3 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (4) | 4 (4)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Diabetic ketosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Haemochromatosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (13) | 12 (15)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 12 (14) | 8 (8)
Hypervolaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 11 (12) | 10 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 11 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (6) | 15 (18)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (5)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Steroid diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8)
Bursal fluid accumulation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibrosis tendinous (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 8 (9) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Necrotising myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 21 (25) | 26 (29)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (2)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4)
Adenocarcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioneuronal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intravascular papillary endothelial hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (6) | 3 (3)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 16 (16)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Metastatic salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 6 (6)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Primary myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (13) | 3 (3)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (4)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Apraxia (Nervous system disorders) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (2) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Basal ganglia stroke (Nervous system disorders) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 8 (9) | 7 (7)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Central nervous system vasculitis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 22 (23) | 25 (27)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 2 (2)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 7 (7)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1)
Embolic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 13 (13) | 7 (7)
Epilepsy (Nervous system disorders) | 3 (3) | 2 (2)
Facial spasm (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 2 (2)
Hepatic encephalopathy (Nervous system disorders) | 3 (3) | 1 (1)
Hypercapnic coma (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 2 (2) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial mass (Nervous system disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 9 (10) | 14 (15)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lateral medullary syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 3 (3) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 6 (7) | 5 (5)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Neurodegenerative disorder (Nervous system disorders) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy chronic (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 4 (4) | 4 (4)
Quadriplegia (Nervous system disorders) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 9 (12) | 2 (2)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Spinal claudication (Nervous system disorders) | 1 (1) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 3 (3) | 4 (4)
Syncope (Nervous system disorders) | 27 (32) | 25 (25)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 8 (8) | 12 (13)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Uraemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0)
Wernicke's encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Peripartum cardiomyopathy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 2 (2) | 1 (1)
Device capturing issue (Product Issues) | 7 (7) | 7 (8)
Device connection issue (Product Issues) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 5 (5) | 7 (7)
Device electrical impedance issue (Product Issues) | 2 (2) | 6 (8)
Device end of service (Product Issues) | 1 (1) | 2 (2)
Device extrusion (Product Issues) | 2 (2) | 0 (0)
Device failure (Product Issues) | 0 (0) | 1 (1)
Device inappropriate shock delivery (Product Issues) | 2 (2) | 1 (1)
Device lead damage (Product Issues) | 8 (8) | 8 (8)
Device lead issue (Product Issues) | 3 (4) | 5 (5)
Device malfunction (Product Issues) | 4 (4) | 4 (4)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Device pacing issue (Product Issues) | 14 (14) | 15 (15)
Device power source issue (Product Issues) | 7 (7) | 7 (7)
Device stimulation issue (Product Issues) | 14 (15) | 27 (28)
Lead dislodgement (Product Issues) | 72 (75) | 53 (61)
Oversensing (Product Issues) | 3 (3) | 3 (3)
Prosthetic cardiac valve malfunction (Product Issues) | 0 (0) | 1 (1)
Stent malfunction (Product Issues) | 1 (1) | 0 (0)
Undersensing (Product Issues) | 1 (1) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment disorder with anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 6 (7)
Delirium tremens (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (4) | 3 (3)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 3 (3) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 10 (10) | 6 (7)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 86 (108) | 84 (95)
Azotaemia (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 7 (9) | 12 (14)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 2 (2)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 10 (12) | 10 (10)
Haematuria (Renal and urinary disorders) | 13 (17) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 4 (4) | 4 (7)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 4 (4) | 4 (6)
Nephropathy (Renal and urinary disorders) | 0 (0) | 2 (2)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 2 (3)
Renal atrophy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal cyst haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 11 (12) | 20 (20)
Renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 2 (5)
Urethral syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 7 (8) | 3 (4)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Breast enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 4 (4)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 5 (8)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 30 (38) | 28 (32)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 7 (11)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cheyne-Stokes respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 28 (35) | 28 (40)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 14 (14)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 19 (24)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 20 (22)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 14 (14)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 27 (28)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Device therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Finger amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Heart valve operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Internal fixation of fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
Intervertebral disc operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 2 (2) | 0 (0)
Medical device implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Mesenteric artery stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Neurostimulator removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Therapeutic procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 6 (6) | 4 (4)
Aortic aneurysm rupture (Vascular disorders) | 2 (2) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 2 (2)
Aortic stenosis (Vascular disorders) | 3 (3) | 9 (10)
Arterial insufficiency (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 2 (2) | 2 (2)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 16 (18) | 20 (20)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 4 (4) | 2 (2)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 18 (22) | 8 (9)
Hypertensive crisis (Vascular disorders) | 5 (5) | 2 (2)
Hypertensive emergency (Vascular disorders) | 3 (3) | 3 (3)
Hypertensive urgency (Vascular disorders) | 9 (9) | 3 (3)
Hypotension (Vascular disorders) | 49 (54) | 54 (64)
Hypotensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 3 (4) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 4 (5) | 1 (1)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Microscopic polyangiitis (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 16 (17) | 11 (12)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Penetrating aortic ulcer (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 24 (34) | 19 (22)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 1 (2)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 2 (3) | 7 (7)
Peripheral vein occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Reperfusion injury (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 3 (3) | 1 (2)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 4 (5)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Superior vena cava stenosis (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 3 (3)
Varicose vein (Vascular disorders) | 1 (1) | 1 (1)
Varicose vein ruptured (Vascular disorders) | 1 (1) | 0 (0)
Vascular stenosis (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | aCRT ON (N=1810) | aCRT OFF (N=1807)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Accelerated idioventricular rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 7 (7) | 5 (5)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 20 (22) | 8 (8)
Angina unstable (Cardiac disorders) | 3 (3) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 5 (5)
Arrhythmia supraventricular (Cardiac disorders) | 5 (5) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 118 (131) | 95 (114)
Atrial flutter (Cardiac disorders) | 8 (8) | 7 (7)
Atrial tachycardia (Cardiac disorders) | 12 (12) | 5 (6)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 3 (3)
Bundle branch block left (Cardiac disorders) | 1 (1) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 179 (236) | 208 (270)
Cardiac failure acute (Cardiac disorders) | 4 (4) | 7 (7)
Cardiac failure chronic (Cardiac disorders) | 10 (10) | 14 (14)
Cardiac failure congestive (Cardiac disorders) | 31 (34) | 32 (38)
Cardiac perforation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac perfusion defect (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 2 (2) | 2 (2)
Cardiomegaly (Cardiac disorders) | 1 (1) | 3 (3)
Cardiomyopathy (Cardiac disorders) | 3 (3) | 3 (4)
Chronic left ventricular failure (Cardiac disorders) | 4 (4) | 7 (7)
Chronotropic incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 3 (3)
Coronary artery disease (Cardiac disorders) | 0 (0) | 4 (4)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 3 (3)
Intrapericardial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 3 (3) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 3 (3)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 1 (1)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 13 (14) | 13 (14)
Pericardial effusion (Cardiac disorders) | 5 (5) | 5 (5)
Pericarditis (Cardiac disorders) | 3 (3) | 0 (0)
Pericarditis constrictive (Cardiac disorders) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 5 (5) | 8 (8)
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 14 (15) | 19 (23)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (5) | 2 (2)
Torsade de pointes (Cardiac disorders) | 1 (1) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 26 (27) | 21 (25)
Ventricular fibrillation (Cardiac disorders) | 7 (8) | 14 (15)
Ventricular tachycardia (Cardiac disorders) | 75 (103) | 81 (126)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Charles Bonnet syndrome (Eye disorders) | 1 (1) | 0 (0)
Ocular ischaemic syndrome (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 4 (4)
Chest pain (General disorders) | 17 (17) | 21 (34)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Decreased activity (General disorders) | 0 (0) | 1 (1)
Device psychogenic complication (General disorders) | 1 (1) | 0 (0)
Drug intolerance (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 9 (9) | 8 (8)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Gravitational oedema (General disorders) | 0 (0) | 1 (1)
Implant site bruising (General disorders) | 3 (3) | 0 (0)
Implant site dehiscence (General disorders) | 3 (3) | 1 (1)
Implant site discharge (General disorders) | 0 (0) | 1 (1)
Implant site erythema (General disorders) | 3 (3) | 0 (0)
Implant site haematoma (General disorders) | 14 (14) | 18 (18)
Implant site haemorrhage (General disorders) | 1 (1) | 1 (1)
Implant site hypoaesthesia (General disorders) | 0 (0) | 2 (2)
Implant site inflammation (General disorders) | 1 (1) | 1 (1)
Implant site oedema (General disorders) | 1 (1) | 0 (0)
Implant site pain (General disorders) | 12 (12) | 14 (14)
Implant site pruritus (General disorders) | 1 (1) | 3 (3)
Implant site rash (General disorders) | 0 (0) | 1 (1)
Implant site swelling (General disorders) | 4 (4) | 3 (3)
Medical device discomfort (General disorders) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 1 (1) | 0 (0)
Medical device site bruise (General disorders) | 1 (1) | 0 (0)
Medical device site discharge (General disorders) | 0 (0) | 1 (1)
Medical device site discomfort (General disorders) | 3 (3) | 0 (0)
Medical device site erosion (General disorders) | 0 (0) | 1 (1)
Medical device site mass (General disorders) | 1 (1) | 0 (0)
Medical device site oedema (General disorders) | 1 (1) | 0 (0)
Medical device site pain (General disorders) | 7 (7) | 4 (4)
Medical device site paraesthesia (General disorders) | 1 (1) | 0 (0)
Medical device site swelling (General disorders) | 1 (1) | 1 (1)
Medical device site vesicles (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3) | 6 (6)
Oedema (General disorders) | 3 (3) | 6 (6)
Oedema peripheral (General disorders) | 27 (30) | 34 (36)
Pacemaker generated arrhythmia (General disorders) | 2 (2) | 0 (0)
Pacemaker syndrome (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 3 (3) | 0 (0)
Phantom shocks (General disorders) | 2 (3) | 4 (4)
Unevaluable event (General disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 3 (3) | 4 (4)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Stitch abscess (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac vein dissection (Injury, poisoning and procedural complications) | 3 (3) | 8 (8)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Device use issue (Injury, poisoning and procedural complications) | 7 (7) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incision site impaired healing (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 4 (4) | 5 (5)
Body fluid analysis (Investigations) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 28 (28) | 12 (12)
Cardiac pacemaker evaluation (Investigations) | 1 (1) | 0 (0)
Carotid bruit (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 2 (2)
Electrocardiogram QRS complex prolonged (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QRS complex shortened (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Electrocardiogram low voltage (Investigations) | 0 (0) | 2 (2)
Heart rate increased (Investigations) | 1 (1) | 1 (1)
Heart rate irregular (Investigations) | 1 (1) | 0 (0)
Heart sounds abnormal (Investigations) | 4 (4) | 4 (4)
Pulmonary arterial pressure increased (Investigations) | 1 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 7 (7) | 11 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 13 (14) | 12 (13)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Electric shock sensation (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Phrenic nerve irritation (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 5 (5)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 10 (10) | 17 (19)
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 6 (6)
Device alarm issue (Product Issues) | 1 (1) | 0 (0)
Device capturing issue (Product Issues) | 7 (8) | 5 (5)
Device deployment issue (Product Issues) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Device electrical impedance issue (Product Issues) | 8 (9) | 7 (9)
Device extrusion (Product Issues) | 0 (0) | 1 (1)
Device inappropriate shock delivery (Product Issues) | 3 (3) | 2 (2)
Device issue (Product Issues) | 1 (1) | 2 (2)
Device lead issue (Product Issues) | 2 (2) | 0 (0)
Device malfunction (Product Issues) | 2 (2) | 2 (2)
Device pacing issue (Product Issues) | 43 (47) | 40 (42)
Device power source issue (Product Issues) | 2 (2) | 1 (1)
Device stimulation issue (Product Issues) | 151 (183) | 153 (192)
Lead dislodgement (Product Issues) | 6 (6) | 3 (3)
Oversensing (Product Issues) | 18 (19) | 26 (30)
Undersensing (Product Issues) | 7 (7) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis interstitial (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 (31) | 28 (28)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Physical assault (Social circumstances) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 2 (3)
Aortic dilatation (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 8 (8) | 11 (11)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Giant cell arteritis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 5 (5) | 0 (0)
Hypertension (Vascular disorders) | 31 (36) | 34 (41)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 41 (43) | 36 (39)
Jugular vein distension (Vascular disorders) | 4 (4) | 4 (4)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Labile blood pressure (Vascular disorders) | 0 (0) | 1 (1)
Labile hypertension (Vascular disorders) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 13 (13) | 10 (11)
Peripheral arterial occlusive disease (Vascular disorders) | 5 (5) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 3 (3) | 0 (0)
Peripheral venous disease (Vascular disorders) | 3 (3) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 2 (2)
Subclavian vein stenosis (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 4 (4)
Superficial vein thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Vascular insufficiency (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Vasoconstriction (Vascular disorders) | 1 (1) | 0 (0)
Vein dissection (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT02205359/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT02205359/SAP_001.pdf